CLINICAL TRIAL: NCT06873737
Title: Analysis of the Levels of HLADR+ Extracellular Vesicles in Women With Preeclampsia as a Early Potential Biomarker
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 4299
Record Dates: First submitted 2025-03-05; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "High risk" (Experimental): Blood sampling from women with high risk to develop preeclampsia in the first, second and third trimester of pregnancy
  Interventions: Other: Blood samples for inflammatory markers
- Low risk (Experimental): Blood sampling from women with low risk to develop preeclampsia in the first, second and third trimester of pregnancy
  Interventions: Other: Blood samples for inflammatory markers

INTERVENTIONS:
Other: Blood samples for inflammatory markers — Blood sampling in the first, second, trimester of pregnancy

SUMMARY:
Analysis of the circulating levels of placenta-derived HLA-DR+ extracellular vesicles in the first, second and third trimester of pregnancy of women with high and low risk to develop preeclampsia.

DETAILED DESCRIPTION:
The aim of this study is to analyze the levels of circulating placenta-derived HLA-DR+ extracellular vesicles in the first, second and third trimester of pregnancy of women with high and low risk to develop preeclampsia to investigate the potential role of HLA-DR as early biomarker.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant Women
* Aged > 18 years

Exclusion Criteria:

* age < 18 years
* women unable to give informed consent
* infectious diseases
* twin pregnancies

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Levels of circulating HLA-DR+ extracellular vesicles | During the first trimester of pregnancy (11-13 weeks +6 days of gestational age), the second trimester (19-22 weeks of gestation) and the third trimester (28-32 weeks of gestation) of pregnancy
  Levels of circulating HLA-DR+ extracellular vesicles during pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Chiara Tersigni, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli, Rome, Italy